CLINICAL TRIAL: NCT02114944
Title: Treatment of Dyspnea in Do-not-intubate (DNI) Patients
Brief Title: Treatment of Dyspnea in Do-not-intubate Patients
Status: Terminated | Type: Observational
Why Stopped: The pandemic shut down study activity and due to personnel problems and retirement of our main collaborator, we were unable to resume afterwards.
Sponsor: Tufts Medical Center (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-11227
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Acute Respiratory Failure; Acute on Chronic Respiratory Failure; Dyspnea
Keywords: Do-not-intubate; DNI; Palliative treatment; Acute respiratory failure; Acute on chronic respiratory failure; Hypoxia; Respiratory acidosis; Hypercarbia; Non invasive ventilation; NIV; CPAP; Oxygen-therapy; High-flow oxygen therapy
MeSH Terms: conditions — Dyspnea; Hypoxia; Acidosis, Respiratory; Hypercapnia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- NIV: Patients with acute respiratory failure or dyspnea and DNI order treated with noninvasive ventilation
  Interventions: Device: NIV; Device: Standard oxygen; Device: HFNC
- CPAP: Patients with dyspnea or acute respiratory failure and DNI order treated with continuous positive airways pressure (CPAP)
  Interventions: Device: CPAP; Device: Standard oxygen; Device: HFNC
- Standard oxygen: Patients with dyspnea and/or acute respiratory failure and DNI order, treated with standard oxygen therapy either via face mask or nasal cannula
  Interventions: Device: Standard oxygen
- HFNC: Patients with dyspnea and/or acute respiratory failure and DNI order treated with high-flow nasal cannula (HFNC).
  Interventions: Device: HFNC

INTERVENTIONS:
Device: NIV — Patients treated, as per attending physician's decision, with noninvasive ventilation
  Groups: NIV
Device: CPAP — Patient treated, as per attending physician's decision, with CPAP
  Groups: CPAP
Device: Standard oxygen — Patient treated, as per attending physician's decision with standard oxygen therapy either as primary respiratory therapy or rest therapy during breaks off CPAP or NIV
  Groups: CPAP; NIV; Standard oxygen
Device: HFNC — Patients treated, as per attending physician's decision, with high-flow nasal cannula either as primary therapy or rest therapy during breaks off NIV or CPAP
  Other Names: High-flow nasal cannula
  Groups: CPAP; HFNC; NIV

SUMMARY:
Patients with severe chronic diseases are often admitted to the hospital complaining of shortness of breath. Some of these patients decide that they do not want placement of a breathing tube in the windpipe to assist their breathing. In this situation, these patients are treated with oxygen, a variety of medications like morphine or masks that are connected to breathing machines, something called bilevel positive airway pressure (BiPAP) or noninvasive ventilation (NIV), to help with their breathing. Not much is known about how much noninvasive ventilation helps these patients, especially how comfortable they feel with it and how much their families think it helps.

Our aim is to monitor use of ways to help breathing in patients who don't want a breathing tube, see how often noninvasive ventilation is used and ask surviving patients, patient's families and caregivers about their experience with noninvasive ventilation and how much it seemed to help.

With our findings, we hope to improve the use of noninvasive ventilation in these patients and come up with ways to relieve their shortness of breath and provide as much comfort as possible.

DETAILED DESCRIPTION:
Background: Respiratory symptoms, dyspnea and acute respiratory failure are often reported in patients admitted to the Hospital with a do-not-intubate (DNI) order. These patients are routinely treated with medical therapy, sometimes to reverse the underlying process, but also often to achieve palliation. The therapies include opioids or anxiolytics, oxygen, CPAP and non-invasive ventilation (NIV) depending on the underlying disease.

Rationale: Considering that most of the available data on the palliative use of NIV are limited to short-term prognosis and are collected selecting DNI patients among those subjects already receiving NIV treatment. A prospective observational study focusing on therapies offered to patients entering the hospital with or switching to a DNI status during the hospitalization would be helpful to fill in the blanks regarding the current palliative treatment of dyspnea in critically ill DNI patients. The assessment of patients' symptoms and comfort and family members' perspective would be important to further understand how the discussion with healthcare proxies and families should be addressed in relation to end-of life-decisions. In addition, the collection of health care providers' impressions on the use of different treatments to alleviate dyspnea and respiratory distress in this situation could help to better understand how to implement palliative treatment of respiratory symptoms in DNI patients.

Our aim is to monitor and establish the prevalence of use of NIV among DNI patients and to assess patients, family members' and caregivers' perspectives on the patient's and their own experience of NIV relative to other approaches to palliating symptoms.

Study design: A prospective, observational study enrolling all consecutive patients with dyspnea and/or acute respiratory failure with DNI orders admitted to the study site.

Study procedures: Subjects participating in the study will be treated as per hospital procedure and according to the attending physician orders, to maintain oxygen saturation at the targeted level and to optimize patient comfort using anxiolytics and narcotics as indicated. No changes in the standard of care will be performed based on participation in the study.

Some data (demographics, medications, vitals, arterial blood gas, history of present illnes and past medical history, treatment plan) will be extracted from medical records. A daily assessment of dyspnea score (Numeric rating scale, (NRS)), comfort (NRS) and pain (NRS) will be performed. Patients and family members will be asked to fill in a questionnaire at day 3. Heal care providers (attending physician, nurse and RT) will be asked to fill in a questionnaire at discharge. Family members and/or patients will be contacted by phone 30 days after discharge to get additional information about patient's outcome.

Research plan: Demographics and baseline characteristics of patients will be summarized for each group overall and by cohorts (DNI on NIV, DNI on CPAP, DNI with no ventilator support). Continuous variables will be reported as mean ± standard deviation. Categorical variables will be reported as n and %. For the primary outcome, a one-way ANOVA will be used to compare the difference in means between the groups. If the data are not normally distributed, the Krusman-Wallis test will be performed. Regression analysis will also be conducted to evaluate the consistency of treatment effects across the cohorts, controlling for potential confounding factors at baseline.

A Chi-square test (or Fisher's exact test if the counts are below 5) will be used to compare the distribution of categorical outcomes between the groups. Where appropriate, generalized linear models will be fitted with categorical and count data to evaluate the consistency of treatment effects across the cohorts, controlling for potential confounding factors at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 or more years of age
* Patients presenting to the study site with dyspnea, respiratory distress and/or acute respiratory failure.
* Patients who have or acquire a DNI order during their hospital stay
* Consent to participate in the study

Exclusion Criteria:

* No exclusion criteria

Termination criteria:

* Withdraw DNI order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to study center will be screened for study entry. Patients with dyspnea and/or acute respiratory failure (regardless the underlying diagnosis) and with a DNI order will be evaluated to define study entry criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of use of Noninvasive ventilation in DNI patients | Day 1

SECONDARY OUTCOMES:
Subjects' comfort | Day 1 to 5
  To define subjects' comfort based on the treatment they are receiving
Dyspnea score | Day 1 to 5
  To define the dyspnea score based on the treatment the subjects are receiving
Family members' impressions | Day 3
  Collect family members' impression on the respiratory device chosen to treat dyspnea and acute respiratory failure
Family member's impressions | Day 30
  Collect family members' impression on the respiratory device chosen to treat dyspnea and acute respiratory failure

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hill, MD, Study Director — Tufts Medical Center
Locations (2):
- Tufts Medical Center, Boston, Massachusetts, United States
- Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Background] Azoulay E, Kouatchet A, Jaber S, Lambert J, Meziani F, Schmidt M, Schnell D, Mortaza S, Conseil M, Tchenio X, Herbecq P, Andrivet P, Guerot E, Lafabrie A, Perbet S, Camous L, Janssen-Langenstein R, Collet F, Messika J, Legriel S, Fabre X, Guisset O, Touati S, Kilani S, Alves M, Mercat A, Similowski T, Papazian L, Meert AP, Chevret S, Schlemmer B, Brochard L, Demoule A. Noninvasive mechanical ventilation in patients having declined tracheal intubation. Intensive Care Med. 2013 Feb;39(2):292-301. doi: 10.1007/s00134-012-2746-2. Epub 2012 Nov 27. PMID 23184037
- [Background] Sinuff T, Cook DJ, Keenan SP, Burns KE, Adhikari NK, Rocker GM, Mehta S, Kacmarek R, Eva K, Hill NS. Noninvasive ventilation for acute respiratory failure near the end of life. Crit Care Med. 2008 Mar;36(3):789-94. doi: 10.1097/CCM.0B013E3181653584. PMID 18209669
- [Background] Nava S, Sturani C, Hartl S, Magni G, Ciontu M, Corrado A, Simonds A; European Respiratory Society Task Force on Ethics and decision-making in end stage lung disease. End-of-life decision-making in respiratory intermediate care units: a European survey. Eur Respir J. 2007 Jul;30(1):156-64. doi: 10.1183/09031936.00128306. PMID 17601972
- [Background] Puntillo K, Nelson JE, Weissman D, Curtis R, Weiss S, Frontera J, Gabriel M, Hays R, Lustbader D, Mosenthal A, Mulkerin C, Ray D, Bassett R, Boss R, Brasel K, Campbell M. Palliative care in the ICU: relief of pain, dyspnea, and thirst--a report from the IPAL-ICU Advisory Board. Intensive Care Med. 2014 Feb;40(2):235-248. doi: 10.1007/s00134-013-3153-z. Epub 2013 Nov 26. PMID 24275901
- [Background] Curtis JR, Cook DJ, Sinuff T, White DB, Hill N, Keenan SP, Benditt JO, Kacmarek R, Kirchhoff KT, Levy MM; Society of Critical Care Medicine Palliative Noninvasive Positive VentilationTask Force. Noninvasive positive pressure ventilation in critical and palliative care settings: understanding the goals of therapy. Crit Care Med. 2007 Mar;35(3):932-9. doi: 10.1097/01.CCM.0000256725.73993.74. PMID 17255876
- [Background] Organized jointly by the American Thoracic Society, the European Respiratory Society, the European Society of Intensive Care Medicine, and the Societe de Reanimation de Langue Francaise, and approved by ATS Board of Directors, December 2000. International Consensus Conferences in Intensive Care Medicine: noninvasive positive pressure ventilation in acute Respiratory failure. Am J Respir Crit Care Med. 2001 Jan;163(1):283-91. doi: 10.1164/ajrccm.163.1.ats1000. No abstract available. PMID 11208659
- [Background] Levy M, Tanios MA, Nelson D, Short K, Senechia A, Vespia J, Hill NS. Outcomes of patients with do-not-intubate orders treated with noninvasive ventilation. Crit Care Med. 2004 Oct;32(10):2002-7. doi: 10.1097/01.ccm.0000142729.07050.c9. PMID 15483407
- [Background] Schettino G, Altobelli N, Kacmarek RM. Noninvasive positive pressure ventilation reverses acute respiratory failure in select "do-not-intubate" patients. Crit Care Med. 2005 Sep;33(9):1976-82. doi: 10.1097/01.ccm.0000178176.51024.82. PMID 16148468
- [Background] Nava S, Ferrer M, Esquinas A, Scala R, Groff P, Cosentini R, Guido D, Lin CH, Cuomo AM, Grassi M. Palliative use of non-invasive ventilation in end-of-life patients with solid tumours: a randomised feasibility trial. Lancet Oncol. 2013 Mar;14(3):219-27. doi: 10.1016/S1470-2045(13)70009-3. Epub 2013 Feb 11. PMID 23406914